CLINICAL TRIAL: NCT04523909
Title: Trajectory of Neuroinflammatory Markers in Cerebrospinal Fluid Prior to and After Thoracic Aortic Surgery: the TURBO Study
Brief Title: Trajectory of Neuroinflammatory Markers in Cerebrospinal Fluid Prior to and After Thoracic Aortic Surgery
Acronym: TURBO
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Wilson F. Abdo, Principal Investigator, Radboud University Medical Center
Other Study IDs: CMO 2017-3774
Record Dates: First submitted 2019-05-06; First posted 2020-08-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction; Thoracic Aortic Aneurysm
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Aortic Aneurysm, Thoracic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — paired blood and CSF samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic aortic surgery patients
  Interventions: Diagnostic Test: Trajectory of neuroinflammatory proteins in CSF and blood

INTERVENTIONS:
Diagnostic Test: Trajectory of neuroinflammatory proteins in CSF and blood — Kinetics of neuroinflammatory markers in CSF and blood

SUMMARY:
Observational prospective pilot study to analyze the trajectory of neuroinflammatory protein expression in cerebrospinal fluid (CSF) in relation to systemic compartment in patients undergoing thoracic aortic surgery.

The aim of this study is to identify and unravel the biochemical (neuroinflammatory) pathways involved in postoperative delirium.

Patient undergoing thoracic aortic surgery will have an external lumbar drain (ELD) in situ on the day before surgery. This ELD remains in place during and three days after surgery to reduce the risk on periprocedural spinal cord ischemia. Paired measurements of CSF and blood will be analyzed.

DETAILED DESCRIPTION:
Major (cardiovascular) surgery is frequently associated with cerebral dysfunction postoperatively. Major surgical procedures account for substantial systemic inflammatory activation. Interestingly, animal models have shown that surgery rather than anaesthetics trigger a neurocognitive decline. An increase of pro-inflammatory cytokines and activation of immune cells mediate this post operative cognitive decline. There is growing support that systemic inflammation can activate the innate immune system of the brain leading to inflammation in the brain ('neuroinflammation'). This neuroinflammation is suggested to play a pivotal role in postoperative delirium and postoperative cognitive decline due to surgery-related systemic inflammation. However little evidence is available on the extend of the neuroinflammation and which biochemical pathways are dysregulated in the brain after surgery.

Thoracic aortic surgery offers the unique opportunity to study the trajectory of protein expression in CSF prior to and after surgery in a non-invasive matter. It is standard of care that an external lumbar drain (ELD) is placed the day prior to surgery and this ELD will remain in place during three postoperative days.

To advance the understanding of the impact of major surgery to the brain, the investigators wish to study the trajectory of protein expression prior to and after thoracic aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Competent patients ≥ 18 years
* Patients who will undergo thoracic aortic surgery and will therefore receive an external lumbar drain as a standard of care procedure.

Exclusion Criteria:

* Patients with meningitis/encephalitis/brain abscess within the last 6 months
* Patients with other neurological conditions: brain injury (acute stroke, brain trauma or cerebral haemorrhage) within the last 3 months, known brain tumours, neurodegenerative disease or known pre-existing cognitive impairment (to a degree that would be compatible with mild cognitive impairment or more).
* Brain or spinal surgery within the last 3 months
* Active infection <2 weeks before surgery
* Patients who object against storage of their body material for scientific reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing thoracic aortic surgery who will therefore receive an external lumbar drain as a standard of care procedure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Trajectory of the concentration of a panel of inflammatory proteins in CSF | 9 timepoints: Baseline (immediately before surgery); Start extracorporeal circulation; Stop extracorporeal circulation (ECC); 2 hours (h) after stop ECC; 4h after stop ECC; 6h after stop ECC; 24h after baseline; 48h after baseline; 72h after baseline
  Changes in CSF cytokine concentrations will be determined (including IL6, IL8, IL10, MCP-1, IL1RA and CX3CL1) between timepoints described below.

SECONDARY OUTCOMES:
Trajectory of the concentration of a panel of inflammatory proteins in plasma | 9 timepoints: Baseline to 72 hours after surgery
  Changes in plasma cytokine concentrations will be determined (including IL6, IL8, IL10, MCP-1, IL1RA and CX3CL1) between timepoints described below.
Trajectory of blood-CSF barrier disruption based on CSF/Plasma albumine ratio | 9 timepoints: Baseline to 72 hours after surgery
  CSF/Plasma albumine ratios will be measured for all timepoints where paired CSF/plasma samples are present
Occurence of postoperative delirium | 14-day incidence of delirium
  Yes or No
Trajectory of brain injury markers in CSF | 9 timepoints: Baseline to 72 hours after surgery
  Changes in brain injury markers will be determined (including NFL, S100B, GFAP, UCHL1, NSE)
Trajectory of brain injury markers in plasma | 9 timepoints: Baseline to 72 hours after surgery
  Changes in brain injury markers will be determined (including S100B, GFAP, UCHL1, NSE)
Changes in ex vivo cytokine production after whole blood stimulation | 5 timepoints: Baseline to 48 hours after surgery
  TNF-a,IL6, IL10
Changes in mHLA-DR expression | 5 timepoints: Baseline to 48 hours after surgery
  monocytic HLA-DR expression assessed by flowcytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Care Medicine, Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided